CLINICAL TRIAL: NCT04041739
Title: The Effect of Fungal Infection on the Outcome Among Diabetic Patients With Foot Osteomyelitis
Brief Title: Fungal Infection in Patients With Diabetic Foot Osteomyelitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rowyda El-sayed Gooda Ali, assistant lecturer, Assiut University
Other Study IDs: fungal diabetic osteomyelitis
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Foot Osteomyelitis
Keywords: fungal infection
MeSH Terms: conditions — Mycoses | interventions — Sensitivity and Specificity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetic foot osteomyelitis: Patients will be subjected to:
  1-History taking including duration of diabetes and ulcer . 2 Clinical examination of ulcer , including diagnosis of osteomyelitis 3- Venous blood will be withdrawn to do the following laboratory tests :
  * HbA1c
  * erythrocyte sedimentation rate(ESR)
  * C reactive protein(CRP)
  * Complete blood culture
  * Serum urea and creatinine 4-culture and sensitivity test 5-Bone fragments and tissue biopsy from infected ulcers 6-Fundus examination
  Interventions: Diagnostic Test: fungal osteomyelitis culture and sensitivity

INTERVENTIONS:
Diagnostic Test: fungal osteomyelitis culture and sensitivity — swabs from ulcer tissue and bone biopsy for culture and sensitivity test and blood sampling

SUMMARY:
estimate the percentage of fungal infection in the pathogenesis of diabetic foot osteomyelitis and assess the outcome of patients with fungal diabetic foot osteomyelitis

DETAILED DESCRIPTION:
Approximately 60% of diabetic foot ulcers (DFUs) are complicated by infection. In more than two-thirds of the cases, infection is the main cause for major lower limb amputation in diabetic patients with foot ulceration. Infections may complicate DFUs in both neuropathic and ischemic ulcers.

However, the simultaneous presence of peripheral arterial disease (PAD) and infection influence the evolution of DFUs, increasing the risk of non-healing and major amputation.

Osteomyelitis is usually due to non-healing ulcers and it is associated with high risk of major amputation.

Osteomyelitis can affect any bone but most frequently the forefoot (90%), followed by the midfoot (5%) and the hindfoot (5%). Forefoot have a better prognosis than midfoot and hindfoot osteomyelitis. Above the ankle amputation risk is significantly higher for hindfoot (50%), than midfoot (18.5%) and forefoot (0.33%).

The diagnosis of osteomyelitis should be first based on clinical signs of infection supported by laboratory, microbiological and radiological evaluation. However, the diagnosis remains a challenge and DFO is often not recognized easily in its initial phase.

Infected wounds usually show purulent secretions or at least two signs of inflammation (swelling, erythema, blood serum secretion or simply blood with or without bone fragments). However, DFO can occur without any local sign of inflammation. Systemic symptoms such as fever and malaise are rare, especially in case of chronic osteomyelitis.

Various clinical findings can help clinicians in detecting bone infection. Two specific clinical signs are predictive of osteomyelitis. The first is the width and depth of the foot ulcer. An ulcer larger than 2 cm2 has a sensitivity of 56% and a specificity of 92%. Deep ulcers (> 3 mm) are more easily associated with an underlying osteomyelitis than superficial ulcers (82% vs 33%).

A second diagnostic criterion to detect DFO is the "probe-to-bone test" (PTB). PBT is performed probing the ulcer area with a sterile blunt probe. If the probe reaches the bone surface the PTB is considered positive. In a study involving 75 diabetic patients, PTB showed a sensitivity of 66%, a specificity of 85% and a positive predictive value of 89%. The same test, evaluated in a subsequent prospective study of 1666 diabetic patients and compared with the culture of infected bones, was found to have a sensitivity of 87%, a specificity of 91%, a positive predictive value of only 57% and a negative predictive value of 98%.

Therefore, in the presence of infected ulcers, a positive PTB test is highly suggestive of osteomyelitis, but a negative test does not exclude it. Instead, in presence of an ulcer without clinical signs of infection, a positive test may be not specific for osteomyelitis while a negative PBT test should exclude a bone infection.

The combination of the PTB test with X-ray improve the sensitivity and specificity in the diagnosis of DFO. Bone infection is also considered in case of visible or exposed bone or discharge of bone fragments.

Diabetic foot osteomyelitis (DFO) is mostly the consequence of a soft tissue infection that spreads into the bone, involving the cortex first and then the marrow. The possible bone involvement should be suspected in all DFUs patients with infection clinical findings, in chronic wounds and in case of ulcer recurrence.The bacterial flora involved has been characterized in much detail and highlights a contemporaneous role for many organisms, both aerobic and anaerobic, in the infective process at a single ulcer site, the metabolic deregulation following DFO may lead to hyperglycemia and a degree of immunocompromise, factors allowing fungi to thrive. In addition, many patients with chronic DFU receive multiple courses of broad-spectrum antibiotics, altering the within wound milieu, suppressing normal flora, and thereby allowing the proliferation of opportunistic pathogens..

Fungal osteomyelitis (OM) is relatively rare. There is scarce literature discussing fungal OM in diabetic foot infections (DFIs).

A role for fungal infection in the pathogenesis of diabetic foot lesions has been suggested previously but remains unstudied

ELIGIBILITY:
Inclusion Criteria:

* All diabetic foot ulcers with osteomyelitis

Exclusion Criteria:

* Patients on corticosteroid therapy.
* Patients on long term antibiotic therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospective cohort study, The study included 100 patients with diabetic foot osteomyelitis.
  They all had long-standing recurrent foot ulceration in which healing had failed despite intensive foot care .
  Ulcer material and bone fragments taken for mycological examination. All ulcers had multiple swabs taken for microbial culture and were examined under direct microscopy .
  Tissue specimens were obtained from the depth of the wound (taking aseptic precautions) after debridement.
  - Venous blood will be withdrawn to do the following laboratory tests :
  * HbA1c
  * erythrocyte sedimentation rate
  * C reactive protein
  * Complete blood culture
  * Serum urea and creatinine 4-culture and sensitivity test 5-Bone fragments and tissue biopsy from infected ulcers 6-Fundus examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
detect magnitude of fungal infection as an etiology causing persistent non healed diabetic foot osteomyelitis | "through study completion, an average of 2 year".
  to evaluate the percentage of fungal infection among foot osteomyelitis and its effect on either healing or amputation.

SECONDARY OUTCOMES:
detect response of healing of resistant infected osteomyelitis to antifungal therapy | 2 years
  to know the impact of adding antifungal treatment may accelerate healing and improve the prognosis.and know the percentage of patients with fungal osteomyelitis healed after antifungal therapy and evaluation of healing response through radiological and laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Haridy, Study Director — Assiut University
Locations (1):
- Assuit University,71511, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Ragnarson Tennvall G, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, van Baal J, van Merode F, Schaper N. High prevalence of ischaemia, infection and serious comorbidity in patients with diabetic foot disease in Europe. Baseline results from the Eurodiale study. Diabetologia. 2007 Jan;50(1):18-25. doi: 10.1007/s00125-006-0491-1. Epub 2006 Nov 9. PMID 17093942
- [Background] Reiber GE, Pecoraro RE, Koepsell TD. Risk factors for amputation in patients with diabetes mellitus. A case-control study. Ann Intern Med. 1992 Jul 15;117(2):97-105. doi: 10.7326/0003-4819-117-2-97. PMID 1605439
- [Background] Nicolau DP, Stein GE. Therapeutic options for diabetic foot infections: a review with an emphasis on tissue penetration characteristics. J Am Podiatr Med Assoc. 2010 Jan-Feb;100(1):52-63. doi: 10.7547/1000052. PMID 20093545
- [Background] Hill SL, Holtzman GI, Buse R. The effects of peripheral vascular disease with osteomyelitis in the diabetic foot. Am J Surg. 1999 Apr;177(4):282-6. doi: 10.1016/s0002-9610(99)00050-1. PMID 10326843
- [Background] Mutluoglu M, Sivrioglu AK, Eroglu M, Uzun G, Turhan V, Ay H, Lipsky BA. The implications of the presence of osteomyelitis on outcomes of infected diabetic foot wounds. Scand J Infect Dis. 2013 Jul;45(7):497-503. doi: 10.3109/00365548.2013.765589. Epub 2013 Feb 5. PMID 23384323
- [Background] Aragon-Sanchez FJ, Cabrera-Galvan JJ, Quintana-Marrero Y, Hernandez-Herrero MJ, Lazaro-Martinez JL, Garcia-Morales E, Beneit-Montesinos JV, Armstrong DG. Outcomes of surgical treatment of diabetic foot osteomyelitis: a series of 185 patients with histopathological confirmation of bone involvement. Diabetologia. 2008 Nov;51(11):1962-70. doi: 10.1007/s00125-008-1131-8. Epub 2008 Aug 22. PMID 18719880
- [Background] Faglia E, Clerici G, Caminiti M, Curci V, Somalvico F. Influence of osteomyelitis location in the foot of diabetic patients with transtibial amputation. Foot Ankle Int. 2013 Feb;34(2):222-7. doi: 10.1177/1071100712467436. Epub 2013 Jan 10. PMID 23413061
- [Background] Eneroth M, Larsson J, Apelqvist J. Deep foot infections in patients with diabetes and foot ulcer: an entity with different characteristics, treatments, and prognosis. J Diabetes Complications. 1999 Sep-Dec;13(5-6):254-63. doi: 10.1016/s1056-8727(99)00065-3. PMID 10764999
- [Background] Lipsky BA. Osteomyelitis of the foot in diabetic patients. Clin Infect Dis. 1997 Dec;25(6):1318-26. doi: 10.1086/516148. PMID 9431370
- [Background] Grayson ML, Gibbons GW, Balogh K, Levin E, Karchmer AW. Probing to bone in infected pedal ulcers. A clinical sign of underlying osteomyelitis in diabetic patients. JAMA. 1995 Mar 1;273(9):721-3. PMID 7853630
- [Background] Lavery LA, Armstrong DG, Peters EJ, Lipsky BA. Probe-to-bone test for diagnosing diabetic foot osteomyelitis: reliable or relic? Diabetes Care. 2007 Feb;30(2):270-4. doi: 10.2337/dc06-1572. PMID 17259493
- [Background] Morales Lozano R, Gonzalez Fernandez ML, Martinez Hernandez D, Beneit Montesinos JV, Guisado Jimenez S, Gonzalez Jurado MA. Validating the probe-to-bone test and other tests for diagnosing chronic osteomyelitis in the diabetic foot. Diabetes Care. 2010 Oct;33(10):2140-5. doi: 10.2337/dc09-2309. Epub 2010 Jul 9. PMID 20622159
- [Background] Aragon-Sanchez J, Lipsky BA, Lazaro-Martinez JL. Diagnosing diabetic foot osteomyelitis: is the combination of probe-to-bone test and plain radiography sufficient for high-risk inpatients? Diabet Med. 2011 Feb;28(2):191-4. doi: 10.1111/j.1464-5491.2010.03150.x. PMID 21219428
- [Background] Alvaro-Afonso FJ, Lazaro-Martinez JL, Aragon-Sanchez J, Garcia-Morales E, Garcia-Alvarez Y, Molines-Barroso RJ. Inter-observer reproducibility of diagnosis of diabetic foot osteomyelitis based on a combination of probe-to-bone test and simple radiography. Diabetes Res Clin Pract. 2014 Jul;105(1):e3-5. doi: 10.1016/j.diabres.2014.04.024. Epub 2014 Apr 28. PMID 24857262
- [Background] Hunt JA. Foot infections in diabetes are rarely due to a single microorganism. Diabet Med. 1992 Oct;9(8):749-52. doi: 10.1111/j.1464-5491.1992.tb01885.x. PMID 1395469